CLINICAL TRIAL: NCT06363396
Title: Fatigue Och Kognitiv Dysfunktion Till följd av Synaptopati Eller Graft Versus Host (GVH) Sjukdom i hjärnan
Brief Title: Fatigue and Cognitive Dysfunction After Allogeneic Stemcell Transplantation, Prospective PET Study
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Ksenia Boriskina, MD, Karolinska Institutet
Other Study IDs: K 2023-7081
Record Dates: First submitted 2024-03-20; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Fatigue; Cognitive Dysfunction
MeSH Terms: conditions — Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples for genotyping for radioligands prior to PET investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with fatigue and cognitive dysfunction: Patients that are one to five years after allogeneic stem cell transplantation and have signs of fatigue and cognitive dysfunction measured by international standarts.
- Patients without fatigue and cognitive dysfunction: Patients that are one to five years after allogeneic stem cell transplantation and have no detectable signs of fatigue and cognitive dysfunction measured by international standarts.

SUMMARY:
This study is the academic study and continuation and further development of a prior project under the leadership of Professor LeBlanc. Patients undergoing allogenic stem cell transplantation are followed up in the outpatient clinic. Here, patients are offered participation the fatigue study measuring both fatigue and cognitive impairment systematically by international standard. Previous study by Boberg et al suggested distinct mRNA and proteomic profiles segregating fatigued from non-fatigued patients as well as patients with or without cognitive impairment. A larger well-defined patient cohort is necessary to confirm these results. Investigators aim to identify specific sets of proteins in the CSF that can serve as potential biomarkers of cognitive dysfunction and/or fatigue. This will be performed with two methods:

* by using mass spectrometry-based proteomics approaches
* Olink technology

PET examinations will be performed on both fatigued and non-fatigued. We will utilize the second generation TSPO radioligand [ 11C]PBR28 as well as the SV2A radioligand [ 11C]UCB-J, both showing high signal-to-noise ratio and adequate test-retest properties.

DETAILED DESCRIPTION:
Investigators plan to enroll 30 patients. Blood and liquor samples will be processed, frozen and stored in biobanks. In addition to the clinical tests we will analyze a large set of proinflammatory cytokines and performed and advanced immunophenotyping to determine the exact signature of immune cells in the blood and and in the liquor. The clinical data after will be systematically analyzed in an uni- and multivariate fashion for underlying risk factors, medications and outcome. This unique set of high quality clinical data together with the results from the lab and the radioimaging will provide a unique data set allowing to answer the research questions associated with the underlying hypothesis.Investigators plan to validate previous findings in a larger cohort and test whether neurocognitive testing battery can predict who will develop fatigue and cognitive dysfunction (CD). We evaluate patients using the Mental Fatigue Scale, Fatigue Severity Scale, and Cambridge Neuropsychological Test Automated Battery (CANTAB) as previously described by our group. Investigators will implement other test batteries (such as GERAS) and evaluate relevance for transplanted patients. Study aims to obtain novel insights into the pathophysiology of fatigue and CD, enabling accurate diagnosis and quantification of the severity. Findings may also be important for other long-term survivors after cancer. The study is expected to generate knowledge on the interaction between immune and synaptic functions which is relevant both for CNS disorders such as MS and Alzheimer's disease but also hematologic malignancies. It ensures the safety of individuals undergoing therapy while successful resolution of complications contributes to the long-term efficacy, promoting sustained health improvement. CANTAB might be directly implemented in the clinic as a tool to evaluate the need for sick-leave and the ability to return to work. Advanced imaging techniques will hopefully become a part of clinical praxis, facilitating the development of targeted interventions.

All patients will perform blood sampling, lumbal puncture, cognitive tests and neuroimaging with PET and MRI.

ELIGIBILITY:
Inclusion Criteria:

* status 1-5 years after HSCT
* no known CNS disorders or psychiatric disturbances

Exclusion Criteria:

* prior TBI or CNS irradiation / intrathecal therapy
* known neurological or psychiatric disorder
* time less then 1 year or over 5 years after transplantation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20-75, both male and female who are 1-5 years after allogeneic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
Results of cognitive tests | 2024-2027
  Measured by CANTAB and Geras panels
Potential biomarkers for fatigue and cognitive dysfunction | 2024-2027
  Measured in blood and csf by using mass spectrometry-based proteomics approaches and Olink technology by selecting different panels of proteins based on data available in the literature.
PET results | 2024-2027
  The primary analysis will focus on the frontal cortex.

SECONDARY OUTCOMES:
Global analyses of the neural connections | 2024-2027
  Global analyses of the neural connections have recently been suggested as potentially important biomarkers of neurocognitive dysfunction after aHSCT

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No